CLINICAL TRIAL: NCT05288660
Title: A Phase 1, Randomized, Blinded, Placebo Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Dose of ALXN1210 Administered Intravenously to Healthy Subjects
Brief Title: A Study of a Single Dose of ALXN1210 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: ALXN1210-HV-101
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: ALXN1210; Pharmacokinetic; Pharmacodynamic; Safety; Immunogenicity
MeSH Terms: interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and on-site medical/nursing staff at the study site were blinded to study drug/dose assignment. The pharmacy staff preparing the investigational products, however, were not blinded to ALXN1210 study drug assignment, but all other site staff, including the Investigator, were blinded. Sponsor staff was unblinded as needed (for example, to participate in the Safety Review Committee and to determine reportability of serious adverse events [AEs]), but was to refrain from sharing any information on study drug assignment with the site staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ALXN1210 200 mg (Experimental): ALXN1210 was administered intravenously.
  Interventions: Drug: ALXN1210
- ALXN1210 400 mg (Experimental): ALXN1210 was administered intravenously.
  Interventions: Drug: ALXN1210
- Placebo (Placebo Comparator): Placebo was administered intravenously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN1210 — All doses of ALXN1210 were administered by IV infusion, using programmable IV infusion pump and IV sets with in-line filters, at a fixed rate of 686 mg/hour (equivalent to 137 milliliters [mL]/hour), excluding interruption for safety or technical reason.
  Other Names: Ultomiris; Ravulizumab
  Arms: ALXN1210 200 mg; ALXN1210 400 mg
Drug: Placebo — All doses of placebo were administered by IV infusion, using programmable IV infusion pump and IV sets with in-line filters, at a fixed rate of 686 mg/hour (equivalent to 137 mL/hour), excluding interruption for safety or technical reason.
  Arms: Placebo

SUMMARY:
This study evaluated the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of a single dose of ALXN1210 in healthy participants, as assessed by electrocardiograms, physical examination, vital signs, laboratory analysis, and assessment of adverse events (AEs).

DETAILED DESCRIPTION:
The participants were randomized in a 2:1 ratio (4 active and 2 placebo) to receive a single dose of ALXN1210 or placebo in the 200-milligram (mg) dose cohort and in a 3:1 ratio (6 active and 2 placebo) to receive a single dose of ALXN1210 or placebo in the 400-mg dose cohort, administered by intravenous (IV) infusion. A 150-day observation period was performed for safety, pharmacokinetic, and pharmacodynamic assessments after study drug administration. Antidrug antibody (ADA) levels were monitored in study participants for the duration of the 150-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index from 18 through 29.9 kilogram (kg)/square meter, inclusive, and weight between 50 and 100 kg, inclusive.
* QT interval (Fridericia's correction); ≤450 milliseconds (msec) for males and ≤470 msec for females at screening and pre-dose on Day 1.
* Willing and able to give written informed consent and comply with the study visit schedule.
* Male participant and his female spouse/partner who was of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (at least 1 of which must be a barrier method), starting at screening and continuing until at least 5 months after the last dose of ALXN1210.
* Documented vaccination with meningococcal conjugate vaccine (MCV4) at least 14 days and not more than 3 years prior to dosing.

Exclusion Criteria:

* Participants in intimate and prolonged contact (defined as living under the same roof or providing personal care) with individuals who are either immunocompromised, or with a specific underlying medical conditions (anatomic or functional asplenia [including sickle cell disease]; congenital complement, properdin, factor D, or primary antibody deficiencies; acquired complement deficiencies [for example, those receiving eculizumab]; and human immunodeficiency virus [HIV]), people younger than 2 years old and older than 65 years old, and professionals exposed to environments of greater risk for meningococcal disease (research, industrial, and clinical laboratory personnel who are routinely exposed to Neisseria meningitidis, military personnel during recruit training [military personnel may be at increased risk when accommodated in close quarters], daycare center workers, or those living on a college or university campus).
* Participants living or working in the Saguenay-Lac-St-Jean area (due to increased incidence of meningococcal infections in that specific area).
* Female participants of childbearing potential, including any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or who was pregnant, breastfeeding, or was not postmenopausal.
* Positive serum pregnancy test at screening or Day -1.
* Serum creatinine greater than the upper limit of normal (ULN) of the testing laboratory at screening and Day -1.
* Alanine aminotransferase or aspartate aminotransferase >ULN of the testing laboratory at screening and Day -1.
* Any of the following hematology tests: hemoglobin <135 grams (g)/L for males and <120 g/L for females; hematocrit <0.41 L/L for males and <0.36 L/L for females; white blood cells <3.5*10^3/microliter (μL) or >ULN of the testing laboratory; absolute neutrophils <1.5*10^3/μL (<1.0*10^3/μL for black race volunteers) or >ULN of the testing laboratory; and platelets <the lower limit of normal of the testing laboratory or >450*10^3/μL at screening and Day -1.
* HIV infection (evidenced by HIV-1 or HIV-2 antibody titer).
* Acute or chronic hepatitis B virus (HBV) infection (evidenced by the presence of HBV surface antigen or immunoglobulin M antibodies against HBV core antigen).
* Acute or chronic hepatitis C virus infection (evidenced by antibody titer).
* Active systemic bacterial, viral, or fungal infection within 14 days prior to dosing.
* Positive QuantiFERON-TB test, indicating possible tuberculosis (TB) infection.
* History of complement deficiency.
* History of malignancy other than basal cell carcinoma.
* Participated in a clinical trial within 30 days before initiation of dosing on Day 1, or used any experimental small-molecule therapy within 30 days prior to dosing on Day 1, or biologic therapy within 90 days prior to initiation of dosing on Day 1 or within 5 half-lives of the product, whichever is greater.
* Major surgery within the last 90 days prior to dosing.
* History of any Neisseria infection; history of unexplained, recurrent infection; or infection requiring treatment with systemic antibiotics within the last 90 days prior to dosing.
* Contraindication to receiving MCV4, including severe (life-threatening) allergic reaction to a previous dose of MCV4; severe (life-threatening) allergy to any vaccine component; previous diagnosis of Guillain-Barré Syndrome.
* History of allergy to excipients of ALXN1210 (that is, polysorbate 80)
* History of allergy to penicillin or cephalosporin, or history of significant allergic reaction to other products (anaphylaxis and angioedema).
* Positive urine drug toxicology screen.
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood of more than 50 mL of blood within 30 days of dosing, or more than 499 mL of blood within 56 days of dosing.
* Clinical diagnosis of any autoimmune or rheumatologic disease (for example, systemic lupus erythematosus, and rheumatoid arthritis) or other condition or medical history that, in the opinion of the Investigator, might interfere with the participant's participation in the study, poses an added risk for the participant, or confounds the assessment of the participant or outcome of the study.
* History of latent or active TB or exposure to endemic areas within 8 weeks prior to the TB test performed at screening.
* Immunization with a live attenuated vaccine 1 month prior to dosing or planned vaccination during the course of the study (except for the vaccination planned by the study protocol).
* Presence of fever (body temperature > 37.6°C) (for example, a fever associated with a symptomatic viral or bacterial infection) within 2 weeks prior to the first dosing.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2015-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Montreal, Canada

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, CSR

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: ALXN1210 200 mg: Participants received single dose of ALXN1210 200 milligrams (mg), via intravenous (IV) infusion on Day 1. Participants were followed up to Day 150.
- Cohort 2: ALXN1210 400 mg: Participants received single dose of ALXN1210 400 mg, via IV infusion on Day 1. Participants were followed up to Day 150.
- Placebo: Participants received placebo matched to ALXN1210 via IV infusion on Day 1. Participants were followed up to Day 150.
Period: Overall Study
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg | Placebo
Started | 4 | 6 | 4
Received at Least 1 Dose of Study Drug | 4 | 6 | 4
Completed | 4 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population was defined as the group of participants who received any dose of the study drug (ALXN1210 or placebo).
Groups:
- ALXN1210 200 mg: Participants received single dose of ALXN1210 200 mg, via IV infusion on Day 1. Participants were followed up to Day 150.
- ALXN1210 400 mg: Participants received single dose of ALXN1210 400 mg, via IV infusion on Day 1. Participants were followed up to Day 150.
- Total: Total of all reporting groups
Arm/Group | ALXN1210 200 mg | ALXN1210 400 mg | Placebo | Total
Number analyzed (Participants) | 4 | 6 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (9.42) | 41.8 (8.33) | 46.3 (8.34) | 43.7 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 2 | 3 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as AEs that occurred on or after the date and time of study drug administration, or those that first occurred before dosing but worsened in frequency or severity after study drug administration. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Day 150
Population: The safety population included the group of participants who received any dose of the study drug (ALXN1210 or placebo).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: ALXN1210 200 mg: Participants received single dose of ALXN1210 200 mg, via IV infusion on Day 1. Participants were followed up to Day 150.
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg | Placebo
Number analyzed (Participants) | 4 | 6 | 4
Participants | 3 | 4 | 4

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of ALXN1210
Description: Blood samples were collected for estimation of Cmax by noncompartmental analyses using Pharsight Knowledgebase Server 4.0.2 and Phoenix WinNonlin 5.3.
Time Frame: Predose, 30 minutes, 4, 8, 24, 48, 96 hours postdose, then at Days 8, 15, 22, 29, 36, 43, 50, 57, 71, 90, 120 and 150
Population: The pharmacokinetic (PK) population included all participants who received ALXN1210 and who had sufficient serum ALXN1210 concentration data to enable the calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (µg/mL)
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg
Number analyzed (Participants) | 4 | 6
microgram/milliliter (µg/mL) | 78.8 (8.02) | 141 (23.9)

3. Secondary Outcome: Time To Maximum Observed Serum Concentration (Tmax) of ALXN1210
Description: Blood samples were collected for estimation of Tmax by noncompartmental analyses using Pharsight Knowledgebase Server 4.0.2 and Phoenix WinNonlin 5.3.
Time Frame: Predose, 30 minutes, 4, 8, 24, 48, 96 hours postdose, then at Days 8, 15, 22, 29, 36, 43, 50, 57, 71, 90, 120 and 150
Population: The PK population included all participants who received ALXN1210 and who had sufficient serum ALXN1210 concentration data to enable the calculation of PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg
Number analyzed (Participants) | 4 | 6
hours | 2.44 [0.800 to 4.248] | 0.657 [0.594 to 1.161]

4. Secondary Outcome: Area Under The Serum Concentration Versus Time Curve From Time Zero To The Time of The Last Quantifiable Concentration (AUC0-t) of ALXN1210
Description: Blood samples were collected for estimation of AUC0-t by noncompartmental analyses using Pharsight Knowledgebase Server 4.0.2 and Phoenix WinNonlin 5.3.
Time Frame: Predose, 30 minutes, 4, 8, 24, 48, 96 hours postdose, then at Days 8, 15, 22, 29, 36, 43, 50, 57, 71, 90, 120 and 150
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microgram*hour/milliliter (µg*hr/mL)
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg
Number analyzed (Participants) | 4 | 6
microgram*hour/milliliter (µg*hr/mL) | 45400 (5240) | 78900 (16300)

5. Secondary Outcome: Area Under The Serum Concentration Versus Time Curve From Time Zero (Dosing) To Infinity (AUCinf) of ALXN1210
Description: Blood samples were collected for estimation of AUCinf by noncompartmental analyses using Pharsight Knowledgebase Server 4.0.2 and Phoenix WinNonlin 5.3.
Time Frame: Predose, 30 minutes, 4, 8, 24, 48, 96 hours postdose, then at Days 8, 15, 22, 29, 36, 43, 50, 57, 71, 90, 120 and 150
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg
Number analyzed (Participants) | 4 | 6
µg*hr/mL | 47600 (6220) | 81900 (17800)

6. Secondary Outcome: Terminal Elimination Rate Constant (λz) of Serum ALXN1210
Description: Blood samples were collected for estimation of λz by noncompartmental analyses using Pharsight Knowledgebase Server 4.0.2 and Phoenix WinNonlin 5.3.
Time Frame: Predose, 30 minutes, 4, 8, 24, 48, 96 hours postdose, then at Days 8, 15, 22, 29, 36, 43, 50, 57, 71, 90, 120 and 150
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg
Number analyzed (Participants) | 4 | 6
1/hour | 0.000900 (0.000146) | 0.000943 (0.0000934)

7. Secondary Outcome: Terminal Elimination Half-life (t½) of Serum ALXN1210
Description: Blood samples were collected for estimation of t½ by noncompartmental analyses using Pharsight Knowledgebase Server 4.0.2 and Phoenix WinNonlin 5.3.
Time Frame: Predose, 30 minutes, 4, 8, 24, 48, 96 hours postdose, then at Days 8, 15, 22, 29, 36, 43, 50, 57, 71, 90, 120 and 150
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg
Number analyzed (Participants) | 4 | 6
days | 32.7 (5.18) | 30.9 (3.20)

8. Secondary Outcome: Total Clearance (CL) of ALXN1210
Description: Blood samples were collected for estimation of CL by noncompartmental analyses using Pharsight Knowledgebase Server 4.0.2 and Phoenix WinNonlin 5.3.
Time Frame: Predose, 30 minutes, 4, 8, 24, 48, 96 hours postdose, then at Days 8, 15, 22, 29, 36, 43, 50, 57, 71, 90, 120 and 150
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliliter/hour
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg
Number analyzed (Participants) | 4 | 6
milliliter/hour | 4.26 (0.620) | 5.06 (0.990)

9. Secondary Outcome: Volume of Distribution (Vd) of ALXN1210
Description: Blood samples were collected for estimation of Vd by noncompartmental analyses using Pharsight Knowledgebase Server 4.0.2 and Phoenix WinNonlin 5.3.
Time Frame: Predose, 30 minutes, 4, 8, 24, 48, 96 hours postdose, then at Days 8, 15, 22, 29, 36, 43, 50, 57, 71, 90, 120 and 150
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg
Number analyzed (Participants) | 4 | 6
milliliters | 4760 (426) | 5340 (727)

10. Secondary Outcome: Percent Change From Baseline in Free Complement Component 5 (C5)
Description: Blood samples were collected for analysis of free C5 concentrations.
Time Frame: Baseline, Day 150
Population: The pharmacodynamic (PD) population consisted of all participants who had sufficient pre and post dose PD assessments (C5 concentration data, chicken red blood cell [cRBC] hemolysis data, classical complement pathway [CCP], complement alternative pathway [CAP], or terminal complement complex [C5b-9]) to enable the evaluation of the PD effects.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg | Placebo
Number analyzed (Participants) | 4 | 6 | 4
percent change | 4.76 (5.52) | 19.88 (12.99) | 24.46 (31.63)

11. Secondary Outcome: Percent Change From Baseline in Total Complement C5
Description: Blood samples were collected for analysis of total C5 concentrations.
Time Frame: Baseline, Day 150
Population: The PD population consisted of all participants who had sufficient pre and post dose PD assessments (C5 concentration data, cRBC hemolysis data, CCP, CAP, or C5b-9) to enable the evaluation of the PD effects.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg | Placebo
Number analyzed (Participants) | 4 | 6 | 4
percent change | 31.02 (8.34) | 23.39 (10.46) | 15.33 (17.86)

12. Secondary Outcome: Percent Change From Baseline in Complement C5b-9
Description: Blood samples were collected for analysis of C5b-9 concentrations.
Time Frame: Baseline, Day 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg | Placebo
Number analyzed (Participants) | 4 | 6 | 4
percent change | -28.22 (19.11) | -40.73 (10.92) | 34.68 (14.61)

13. Secondary Outcome: Percent Change From Baseline in Chicken Red Blood Cell Hemolysis
Description: Blood samples were collected for analysis of cRBC hemolysis.
Time Frame: Baseline, Day 150
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg | Placebo
Number analyzed (Participants) | 4 | 6 | 4
percent change | 9.86 (7.57) | 15.30 (29.35) | -4.68 (4.76)

14. Secondary Outcome: Percent Change From Baseline In Complement Classical Pathway (CCP) Activity
Description: Blood samples were collected for analysis of CCP.
Time Frame: Baseline, Day 150
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg | Placebo
Number analyzed (Participants) | 4 | 6 | 4
percent change | -13.16 (13.65) | 5.34 (6.05) | -1.81 (10.95)

15. Secondary Outcome: Percent Change From Baseline In Complement Alternative Pathway (CAP) Activity
Description: Blood samples were collected for analysis of CAP.
Time Frame: Baseline, Day 150
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg | Placebo
Number analyzed (Participants) | 4 | 6 | 4
percent change | -23.61 (19.91) | -24.66 (18.48) | -22.08 (13.18)

16. Secondary Outcome: Percentage of Participants With Positive Anti-Drug Antibody (ADA)
Description: Blood samples were collected to evaluate antibody response through development of ADAs.
Time Frame: Baseline up to Day 150
Population: The immunogenicity analysis population consisted of all participants who had pre-dose and at least one post-dose human anti-human antibodies (HAHA) sample collected. The outcome measure was planned to be analyzed for Cohort 1: ALXN1210 200 mg and Cohort 2: ALXN1210 400 mg arms only.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: ALXN1210 200 mg | Cohort 2: ALXN1210 400 mg
Number analyzed (Participants) | 4 | 6
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 150
Description: The safety population was defined as the group of participants who received any dose of the study drug (ALXN1210 or placebo).
Arm/Group | ALXN1210 200 mg | ALXN1210 400 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 4/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN1210 200 mg (N=4) | ALXN1210 400 mg (N=6) | Placebo (N=4)
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN1210 200 mg (N=4) | ALXN1210 400 mg (N=6) | Placebo (N=4)
Headache (Nervous system disorders) | 0 | 3 | 3
Presyncope (Nervous system disorders) | 0 | 0 | 1
Infusion Site Pain (General disorders) | 1 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1
Chest Pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1
Feeling Hot (General disorders) | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 1
Neutrophil Count Decreased (Investigations) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Metal Fume Fever (Injury, poisoning and procedural complications) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 1
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes